CLINICAL TRIAL: NCT06354777
Title: REView of ProcEdural FactoRs and Outcomes After Atrial Fibrillation Ablation With Active Esophageal COOLing: A Sub-study of the REAL AF Registry
Acronym: EVERCOOL AF
Status: Active, not recruiting | Type: Observational
Sponsor: Heart Rhythm Clinical and Research Solutions, LLC (Other)
Collaborators: Attune Medical (Other)
Responsible Party: Sponsor
Other Study IDs: EVERCOOL AF
Record Dates: First submitted 2024-02-28; First posted 2024-04-09 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Subjects who undergo left atrial ablation using esophogeal cooling: Study population will consist of consecutive male and female patients in the REAL AF Registry who have symptomatic Paroxysmal Atrial Fibrillation (PAF) or Persistent Atrial Fibrillation (PsAF) and undergo left atrial ablation with active esophageal cooling for the treatment of atrial fibrillation.
  Interventions: Device: Atrial Ablation

INTERVENTIONS:
Device: Atrial Ablation — Left atrial radiofrequency ablation for the treatment of atrial fibrillation; this may include Pulmonary Vein Isolation (PVI) with or without additional ablation lesions as warranted during the procedure

SUMMARY:
This is a multi-center sub-study examining the effectiveness of active esophageal cooling on subjects undergoing left atrial ablation for symptomatic Paroxysmal Atrial Fibrillation or Persistent Atrial Fibrillation.

DETAILED DESCRIPTION:
Treatment of atrial fibrillation, using pulmonary vein isolation, involves some risks to collateral structure, including the esophagus. Active esophageal cooling has shown benefits in multiple studies when used in the treatment of Paroxysmal Atrial Fibrillation or Persistent Atrial Fibrillation during left atrial ablation. The largest randomized, controlled trial to date, the IMPACT study, found an 83% reduction in endoscopically identified esophageal lesions when using the active cooling, with a dedicated device, compared to standard esophageal monitoring, with no difference in Atrial Fibrillation recurrence rates at follow-up. Recent analyses have suggested additional effects from active esophageal cooling during pulmonary vein isolation, including reductions in procedure time, reductions in fluoroscopy usage, reductions in post-ablation discomfort, and improvements in long-term freedom from arrhythmia. Further investigation of these associations is important to better understand the magnitude of these findings in a variety of clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic Paroxysmal Atrial Fibrillation (AF episode terminate spontaneously within 7 days) or Persistent Atrial Fibrillation (AF sustained beyond 7 days) who, in the opinion of the investigator, are scheduled for ablation for Atrial Fibrillation with active esophageal cooling.
* >18 years of age
* Index or redo ablation procedure and enrolled in the REAL AF Registry
* Willing and able to provide informed consent and complete GERD questionnaire.

Exclusion Criteria:

* For the purpose of this sub-study, candidates will be excluded if they meet any of the following criteria:
* Enrolled in an investigational drug or device clinical trial, or any trial that dictates the treatment plan.
* In the opinion of the investigator, any known contraindication to an ablation procedure.
* <18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sub-study will consist of consecutive male and female patients enrolled in the REAL AF Registry who have symptomatic Paroxysmal Atrial Fibrillation (PAF) or Persistent Atrial Fibrillation (PsAF) and undergo left atrial ablation for the treatment of atrial fibrillation.
Sampling Method: Probability Sample
Enrollment: 312 (Actual)
Dates: Start 2024-04-03 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
To measure procedural efficacy after atrial fibrillation ablation in patients treated with active esophageal cooling. | 90 days
  Freedom from atrial arrhythmia recurrence at 90 days post procedure.
To measure procedural efficacy after atrial fibrillation ablation in patients treated with active esophageal cooling. | 12 months
  Freedom from atrial arrhythmia recurrence at 12 months post procedure
To measure long term safety after atrial fibrillation in patients treated with active esophageal cooling. | up to 12-months
  Adverse events from post-procedure through the 12-month office visit date
Patient reported outcomes in patients treated with active esophageal cooling. | 7-14 days
  Outcomes reported in modified Gastroesophageal Reflux Disease (GERD) questionnaire. Scale will be scored from "0" (no symptoms) to "3" (maximum symptoms). Higher scores indicate a worse outcome.
Physician reported outcome post procedure with active esophageal cooling. | Up to 2 months
  Assessed using Physician Survey Questionnaire of multiple-choice questions.

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Sharkoski, MPH, Study Chair — Haemonetics Corporation
Locations (6):
- United States (6):
  - Valley Heart Rhythm Specialists, Chandler, Arizona
  - Ascension St. Vincent Hospital Indianapolis, Indianapolis, Indiana
  - Corewell Health Research Institute, Royal Oak, Michigan
  - Christ Hospital, Cincinnati, Ohio
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - MultiCare Institute for Research & Innovation, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No